CLINICAL TRIAL: NCT04078087
Title: The Effect of Body Mass Index In Relation To Menstrual Cycle Phase on Propofol Injection Pain
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Raham Hasan Mostafa, MD, Assistant Professor of Anesthesia, Ain Shams University
Other Study IDs: R43/2019; R43/2019 (Registry Identifier: Ain Shams research ethical committee)
Record Dates: First submitted 2019-09-02; First posted 2019-09-04 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Injection Site Coldness; Propofol Adverse Reaction
Keywords: Body mass index; Follicular phase; Injection pain; Luteal phase; Menopause; Menstrual cycle; Visual analogue scale
MeSH Terms: interventions — Adiposity; O-antigen, Acinetobacter strain 90

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non obese: Non obese (whether normal weight or overweight) = Group "NO"
  Interventions: Drug: Non obese
- Obese: obese = Group "O"
  Interventions: Drug: Obese.

INTERVENTIONS:
Drug: Non obese — After standard anesthesia monitoring, Administration of oxygen was performed for 3 minutes with 10 L/min fresh gas flow of 100% oxygen. After oxygen administration, 25% of (2 mg/kg) total propofol dose was injected over 3-5 seconds (Propofol Lipuro 1%, B. Braun Melsungen AG, Germany). The patients were observed and asked immediately whether they had pain in the arm, its VAS score, type of pain (burning, parathesia or other) and its onset was documented (to differentiate early or late type of pain).
  Other Names: Group NO
  Groups: Non obese
Drug: Obese. — After standard anesthesia monitoring, Administration of oxygen was performed for 3 minutes with 10 L/min fresh gas flow of 100% oxygen. After oxygen administration, 25% of (2 mg/kg) total propofol dose was injected over 3-5 seconds (Propofol Lipuro 1%, B. Braun Melsungen AG, Germany). The patients were observed and asked immediately whether they had pain in the arm, its VAS score, type of pain (burning, parathesia or other) and its onset was documented (to differentiate early or late type of pain).
  Other Names: Group O
  Groups: Obese

SUMMARY:
There are suggestions from experimental pain studies that pain perception in patients with severe obesity differs compared with individuals with lower BMI values, with a tendency for patients with severe obesity to be hypoalgesic - that is, to have reduced numerical pain scores to a variety of painful stimuli. That finding could be related to: associated reduced cognitive function (complex attention, verbal and visual memory, and decision making) in severe obesity.

The purpose of this study is to determine differences between females' pain levels whether they are obese or non-obese, during different menstrual phases (premenstrual, postmenstrual and menopausal phases) through propofol injection pain given for induction of GA

DETAILED DESCRIPTION:
* Study population Ninety patients, 18 years - 65yor older, physical status ASA I&II, scheduled to undergo elective gynecological surgery, will be enrolled in this prospective observational study.
* Patients' recruitment Patients will be recruited after admission to the hospital, same day they scheduled for surgery. All women who will meet inclusion criteria and gave written informed consent for participation in the study will be enrolled.

Patients will be divided into 2 groups according to BMI levels: Non obese (whether normal weight or overweight) = Group "NO" and obese = Group "O". Normal weight is defined as BMI 18.5-24.9, overweight as BMI 25.0-29.9 and obesity as BMI ≥ 30. [8] This study is a single blind study, where patients are aware of their menstrual status but supporting examiner is not aware of the patients' menstrual status.

Patients will be instructed on a vertical VAS 0-10 cm where (0) is marked as no pain and (10) is marked as the worst pain ever felt After standard anesthesia monitoring, Administration of oxygen will be performed for 3 minutes with 10 L/min fresh gas flow of 100% oxygen. After oxygen administration, 25% of (2 mg/kg) total propofol dose will be injected over 3-5 seconds (Propofol Lipuro 1%, B. Braun Melsungen AG, Germany). The patients will be observed and asked immediately whether they had pain in the arm, its VAS score, type of pain (burning, parathesia or other) and its onset will be documented (to differentiate early or late type of pain).

Another anesthesiologist, who is unaware of the study groups, will assess the intensity of pain after propofol injections.

ELIGIBILITY:
Inclusion Criteria:

* 18 years - 65yor older,
* physical status ASA I&II

Exclusion Criteria:

* irregular menstrual cycle,
* those who received hormonal therapy for any cause,
* on oral contraceptive pills,
* breast feeding,
* pregnant,
* history of total abdominal hysterectomy and/or bilateral salphingo-opherectomy.
* patients who had difficulty in understanding the visual analogue scale (VAS)/ pain scoring systems,
* renal or hepatic insufficiency,
* anticipated difficult tracheal intubation, and
* hypersensitivity to the study drugs.
* Also, patients on antidepressants and analgesics

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Study Population: 18 years - 65yor older, physical status ASA I&II, scheduled to undergo elective surgery, were enrolled in this prospective observational study
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
VAS score | immediately after injection
  Incidence & severity of propofol injection pain (Mild pain was defined as VAS score 0-3, Moderate as VAS score 4-6, Severe as VAS score 7-10).

SECONDARY OUTCOMES:
Type of Propofol injection pain, early or late (after 10 seconds) | after 10 seconds
  Type of Propofol injection pain, early or late (after 10 seconds)
Hemodynamic variables | till 5 minutes after tracheal intubation
  Hemodynamic variables were recorded before administration of the IV anesthetic, as well as after TI and 5 minutes later
Rate pressure products | till 5 minutes after tracheal intubation
  Rate pressure products were calculated (an indicator of the heart's demand for oxygen) at same hemodynamic predetermined measuring timings.

CONTACTS AND LOCATIONS:
Overall Officials: Raham H Mostafa, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Excel Sheet, individual deidentified participant data will be shared study protocol, statistical analysis plan will be shared